CLINICAL TRIAL: NCT06594016
Title: Expanded Access to Fosigotifator
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-10780; C25-693 (Other: Abbvie)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Vanishing White Matter; Cree Leukoencephalopathy
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme; Fosigotifator; FGT; ABBV-CLS-7262; 2025-10780; C25-693; Vanishing White Matter; Cree Leukoencephalopathy
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Fosigotifator — Oral
  Other Names: FGT; ABBV-CLS-7262

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to Fosigotifator prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=2025-10780